CLINICAL TRIAL: NCT05200962
Title: Investigating the Mechanism of Action of Electrical Brain Stimulation for Cognitive Impairment in Schizophrenia: a tDCS-fMRI Study
Brief Title: Electrical Brain Stimulation for Cognitive Impairment in Schizophrenia: a tDCS-fMRI Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: University of British Columbia (Other); Ruhr University of Bochum (Other); Leibniz Research Centre for Working Environment and Human Factors (Other); University of Tehran (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021_01_GF16
Record Dates: First submitted 2021-12-22; First posted 2022-01-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Cognitive Impairment
Keywords: Schizophrenia; cognitive impairment; Transcranial direct current stimulation; fMRI
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS group (Experimental): The experimental arm receives real (or active) electrical stimulation for 20 minutes
  Interventions: Device: transcranial direct current stimulation
- sham tDCS group (Sham Comparator): The sham arm receives sham (or no real) intervention in which stimulation lasts for 30 seconds and ends afterward.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — In tDCS, direct electrical currents are generated by an electrical stimulator and are noninvasively delivered to the scalp through a pair of saline-soaked sponge electrodes (7×5 cm).
  Other Names: tDCS; tES

SUMMARY:
The purpose of this study is to investigate the mechanism of action of transcranial electrical brain stimulation over the dorsolateral prefrontal cortex for cognitive impairment in schizophrenia. To do so the effect of a 3-mA stimulation protocol on neurocognitive functions will be investigated using behavioral performance and fMRI.

DETAILED DESCRIPTION:
Thirty schizophrenic patients will be recruited after meeting the inclusion criteria and will be randomly assigned to active and sham stimulation groups. A single session of concurrent prefrontal tDCS/fMRI will be conducted. Participants will undergo baseline task performance before the intervention. One week later, they will undergo the tDCS intervention (active or sham) next to the scanner during which they perform the working memory task varying in cognitive load. They will perform the task 24 h later again. They will be then transferred to MRI scanner right after stimulation

ELIGIBILITY:
Inclusion Criteria:

* men or women (18-50 yrs old) with a DSM 5 SCZ diagnosis,
* If female, negative urine pregnancy test
* significant cognitive impairment (1 SD below the norm on the working memory/executive functioning task performance)
* feasibility for tDCS interventions according to safety guidelines
* stable medication regime especially the classical neuroleptics and all CNS-activating medications, if taken, 4-6 weeks before the experiment
* fluency in the native language
* right-handed
* ability to provide informed consent.

Exclusion Criteria:

* pregnancy
* alcohol or substance dependence
* history of seizure
* history of neurological disorder
* history of head injury
* Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces). Eligibility will be determined by the "MRI Safety Screening Questionnaire" and verified, if necessary, by a radiology consultant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Working memory behavioral performance | up to 24 hours after the intervention
  A computerized version of 3- back letter task, optimized for administration in a functional MRI environment will be employed during the experiment
Modifications to blood-oxygen-level-dependent (BOLD) signal | up to 1 hour
  Changes to blood-oxygen-level-dependent (BOLD) signal (arbitrary units) of brain areas that are implicated in cognitive impairment and pathophysiology of schizophrenia during the working memory task, as measured by fMRI following the intervention between the active and sham groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The National Brain Mapping Laboratory (NBML), Tehran, Iran

IPD SHARING:
Plan to Share IPD: No